CLINICAL TRIAL: NCT00835913
Title: Autonomic Nervous System Alteration Induce by Sepsis:Assessment and Prognosis Impact
Brief Title: Autonomic Nervous System Alteration Induce by Sepsis: Assessment and Prognosis Impact
Acronym: SNA&Sepsis
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 06PHR04; 2008-A00453-52
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2010-07

CONDITIONS: Septic Shock; Severe Sepsis
Keywords: Autonomic nervous system; Sepsis shock; severe sepsis; sinusal change; Myocardiac fixing; NTproBNP; Patient in intensive care unit with sepsis shock or severe; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peptid and protein sAmple
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Severe sepsis and septic shock are causes of admission in intensive care units.Modification of natriuretic peptid including NT-proBNP and cardiac autonomic nervous system alteration are reported in sepsis shock and severe sepsis and seems to link to patient prognosis admitted to intensive care units.

DETAILED DESCRIPTION:
Our principal aim is to characterize modulation of cardiac sympathic nervous system in sepsis through the study of sinusal change and myocardiac fixing of MIBG.

The second aim is 1)to assess links between alteration of cardiac sympathic nervous system and NT-PRoBNP variations in sepsis and 2)To know prognostic impact in sympathic nervous system compare to NTproBNP.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years admitted in intensive care unit and having severe sepsis criteria or septic shock documented or suspected define as Bone Criteria
* hemodynamically stable situation
* sinusal rhythm
* Patient for social security

Exclusion Criteria:

* Minors
* Patient under guardianship or trusteeship
* pregnant or lactating women
* diabetic
* cardiomyopathy known and/or treated or detect in admission
* electro-systolic process permanent or transitory
* neurological history or degenerative pathology
* chronic respiratory insufficiency
* Chronic renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patient transfer in intensive care unit with sepsis chock or severe sepsis define as Bone criteria.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Sinusal variability analysis and myocardic fixation of MIBG performed in 48 hours post admission | 48 hours post admission

SECONDARY OUTCOMES:
plasmatic measure of NT-ProBNP and catecholamine at admission, day 2 and last day of hospitalisation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: SCHWEBEL Carole, PH, Principal Investigator — Unit intensive care
Locations (1):
- University Hospital Grenoble, Grenoble, France